CLINICAL TRIAL: NCT02251860
Title: A Prospective, Non-Interventional Study in Germany to Evaluate the Long-Term Effectiveness and Tolerability of Subcutaneously Administered RoActemra® (Tocilizumab; TCZ) in Patients With Rheumatoid Arthritis in Daily Clinical Practice (as Recommended in Label)
Brief Title: Study of Tocilizumab (RoActemre) Administered Subcutaneously in Participants With Rheumatoid Arthritis in Everyday Clinical Practice
Acronym: ARATA
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29087
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with Rheumatoid Arthritis: Participants with active rheumatoid arthritis who are prescribed tocilizumab treatment according to the marketing authorization by their physician will be followed under routine conditions over an observation period of up to 2 years if baseline and disease characteristics data are available.

SUMMARY:
ARATA is a prospective, non-interventional, multicenter, observational study in Germany to evaluate the long-term effectiveness and tolerability of subcutaneously administered tocilizumab in participants with rheumatoid arthritis in daily clinical practice. Participants will be followed over an observation period of up to 2 years after the initial injection.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have not yet been treated with tocilizumab
* Participants who have received the first injection with tocilizumab maximum 1 month before inclusion in the study and the necessary baseline data and disease characteristics are present

Exclusion Criteria:

* Participants who at the time of the study inclusion are participating in a different interventional study on rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with active rheumatoid arthritis who are prescribed subcutaneous tocilizumab treatment by their physician prior to and independent of the inclusion of the participant into the study. Participant can be enrolled into the study at maximum 1 month after first tocilizumab administration if baseline and disease characteristics data are available.
Sampling Method: Non-Probability Sample
Enrollment: 1454 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission Defined by Disease Activity Score based on 28 Joints-Erythrocyte Sedimentation Rate (DAS28-ESR) in Participants with Previous Biological Disease Modifying Anti-Rheumatic Drug (bDMARD) Treatment | Up to Week 104
Percentage of Participants with Clinical Remission Defined by DAS28-ESR in bDMARD Naïve Participants | Up to Week 104

SECONDARY OUTCOMES:
Change from Baseline in Mean DAS28-ESR Score | Baseline up to Week 104
Percentage of Participants with Continuation of Tocilizumab | Up to Week 104
Mean Retention Time of Tocilizumab | Up to Week 104
Percentage of Participants with Adverse Events (AEs) During Tocilizumab Treatment | From Baseline up to tocilizumab treatment discontinuation (Up to Week 104)
Percentage of Participants with Concomitant Treatment with Methotrexate (MTX) | Up to Week 104
Percentage of Participants with Low Disease Activity Defined by DAS28-ESR | Up to Week 104
Percentage of Participants with Clinical Remission Defined by Clinical Disease Activity Index (CDAI) | Up to Week 104
Percentage of Participants with Low Disease Activity Defined by CDAI | Up to Week 104
Change from Baseline in Mean CDAI Score | Baseline up to Week 104
Percentage of Participants with Critical Difference Related to DAS28 (Dcrit)-Response | At Month 3 and Month 6
Percentage of Participants with Concomitant Treatment with Glucocorticoids (GCs) | Up to Week 104
Mean Dose Used for Concomitant GCs | Up to Week 104
Percentage of Participants with Dose Reduction for Concomitant GCs | Up to Week 104
Treatment Satisfaction Visual Analogue Scale (VAS) | Up to Week 104
Treatment User-Friendliness VAS | Up to Week 104
Percentage of Participants with Treatment Adherence | Up to Week 104
Response to Follow-up Treatment in Case of Switch from Tocilizumab | Up to Week 104
Percentage of Participants with Adverse Events During Follow-up Treatment | Up to Week 104
Health Assessment Questionnaire-Disability Index (HAQ-DI) Score | Up to Week 104
Hannover Functional Ability Questionnaire (FFbH) Score | Up to Week 104
Percentage of Participants by Type of Physical Exercise | Up to Week 104
Percentage of Participants by Frequency of Physical Exercise | Up to Week 104
Percentage of Participants by Duration of Physical Exercise | Up to Week 104
Fatigue-VAS | Up to Week 104
Sleep Disturbance-VAS | Up to Week 104
State-Trait Anxiety Inventory (STAI) Questionnaire | Up to Week 104
Beck Depression Inventory (BDI) Questionnaire | Up to Week 104
Work Productivity and Activity Impairment Questionnaire: Rheumatoid Arthritis (WPAI-RA) | Up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- CIRI - Centrum für Innovative Diagnostik und Therapie Rheumatologie/ Immunologie (GmbH), Frankfurt, Germany